CLINICAL TRIAL: NCT06936423
Title: Exploring Efficacy and Safety: A Comparative Prospective Cohort Study Of Needlescopic Inguinal Hernia Repair Versus Open Herniotomy In Pediatrics
Brief Title: Comparative Study of Needlescopic Inguinal Hernia Repair Versus Open Herniotomy
Acronym: Needlescopic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No.IRB 00006379
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2024-01

CONDITIONS: Indirect Inguinal Hernia; Pediatric
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open herniotomy Group (Active Comparator)
  Interventions: Procedure: Open herniotomy
- Needlescopic percutaneous Internal Ring Suturing group (Active Comparator)
  Interventions: Procedure: Needlescopic percutaneous Internal ring suturing

INTERVENTIONS:
Procedure: Open herniotomy — Open inguinal herniotomy through inguinal incision then dissection and separation/ligation of the hernial sac
  Arms: Open herniotomy Group
Procedure: Needlescopic percutaneous Internal ring suturing — Laparoscopic extracorporeal percutaneous Internal ring suturing using epidural needle and prolene/ethibond suture
  Arms: Needlescopic percutaneous Internal Ring Suturing group

SUMMARY:
This study aims to compare between two techniques to treat hernia in children which are Needlescopic inguinal hernia repair and Open classic surgery as regard operative time, cosmetic appearance, recurrence and other complications

DETAILED DESCRIPTION:
Study Procedures:

Preoperative assessment :

1. Detailed history including age, sex, complain (groin swelling increasing in size with cough and crying) and past surgical and medical history.
2. General and local examination including reducible swelling forwards, upwards and laterally (inguinoscrotal in males and inguinal in females). If any sign or symptoms of irreducibility or strangulation present (abdominal distention, vomiting, constipation, tense, tender or erythematous inguinal swelling) patient should be excluded.
3. Investigations: Inguinal ultrasound is only done in cases of query history or uncertain examination or to exclude bilateral pathology.
4. Preoperative preparation included complete blood count, coagulation profile and complete fasting hours.

Operative technique:

Anaesthesia: General anaesthesia using endotracheal intubation and muscle relaxant plus local anaesthesia in the form of caudal block.

Position: supine. Sterilization of operative field from Xiphisternal joint to mid-thigh by Povidone-iodine solution.

Operative steps:

A) Needlescopic Internal Ring Suturing with Epidural needle.

EQUIPMENT/SUTURE:

1. One 5-mm trocar and 5-mm lens 30° or 0° laparoscopy.
2. Epidural needle.
3. Prolene 2-0 suture.

STEPS:

1. A 5mm port for the camera is introduced at umbilicus.
2. Hydrostatic dissection of the peritoneum of the cord structures is done by injecting saline in males.
3. The suture is introduced through the barrel of the epidural needle.
4. Maintaining both ends of the preloaded suture extra peritoneal, the needle is advanced under the peritoneum around lateral half of the internal ring.
5. The peritoneum is entered and the suture advanced into the abdominal cavity, creating a loop.
6. The needle is removed, leaving the loop in place.
7. The needle is entered again through the same skin puncture site around the medial half of the ring and enter the peritoneum, leaving a small space above the vas deferens and testicular vessels to prevent injury.
8. The loop of suture is introduced into the hollow of the needle again and advance the suture into the first loop.
9. Withdraw the needle.
10. Catch the suture end in the loop and withdraw them together then the suture is tied extra corporeally.

B) Open surgery repair:

1. Groin incision.
2. Dissecting the hernia sac from the spermatic cord in males.
3. Suture tightening of the hernia sac base. The Patients will be discharged after 4 hours post-operative.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female patients. 2. Age between 4 to 12 years. 3. Bilateral or unilateral indirect inguinal hernia

Exclusion Criteria:

* 1. Age below 4 year and above 12 years. 2. Irreducible inguinal hernia. 3. Recurrent inguinal hernia. 4. Patient not fit for Laparoscopic Surgery. 5. Direct inguinal hernia. 6. Sliding type of indirect inguinal hernia. 7. Double pathology like associated undescended testis, vaginal hydrocele, encysted hydrocele and hydrocele of canal of Nuck.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Intraoperative outcomes | From the start of anesthesia till the end of operation
  Operative time. / Intraoperative complication. / Rate of conversion to open surgery.
1st Post-operative visit | After 1 week post operative
  for removal of wound dressing and assessment of wound for infection if present or recurrence.
2nd post-operative visit | After 1 month post operative
  For assessment of : Cosmetic appearance. Recurrence. Hydrocele if present
3rd post-operative visit | After 3 month post operative
  tfor assessment of : Cosmetic appearance. Recurrence. Hydrocele

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared once study is completed
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Before may 2025
Access Criteria: Free